CLINICAL TRIAL: NCT01807663
Title: Validation of a Dynamic Evaluation Tool in Respiratory Failure by Ambulatory Inductance Plethysmography
Brief Title: Validation of a Dynamic Evaluation Tool in Respiratory Failure
Acronym: TELERESP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Healthy volonteers study results show that the device is not enough reliable
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Collaborators: Adep Assistance (Other)
Responsible Party: Principal Investigator, david orlikowski, MDPHD, Centre d'Investigation Clinique et Technologique 805
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-A01280-43
Record Dates: First submitted 2013-02-26; First posted 2013-03-08 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Respiratory Failure
Keywords: neuromuscular disease
MeSH Terms: conditions — Respiratory Insufficiency; Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- healthy volunteers (Experimental): Free breath monitoring. Correlation between two device for recording parameters of ventilation.
  Interventions: Device: healthy volonteers; Device: Free breath monitoring
- Chronic patient (Experimental): Free breath monitoring. Number of pathological respiratory events (apneas, hypopneas, paradoxical breath) compared with the recording of the PtCO2 and the SpO2)
  Interventions: Device: healthy volonteers; Device: Free breath monitoring
- ACUTE PATIENT (Experimental): Free breath monitoring. Number of pathological respiratory events (apneas, hypopneas, paradoxical breath) compared with the recording of the PtCO2 and the SpO2)
  Interventions: Device: healthy volonteers; Device: Free breath monitoring

INTERVENTIONS:
Device: healthy volonteers — Monitoring respiratory function of both acute and chronic neuromuscular patients during weaning or free breath period.
  Other Names: Visuresp system : wireless inductance plethysmography system
Device: Free breath monitoring — Monitoring respiratory function of both acute and chronic neuromuscular patients during weaning or free breath period.
  Other Names: Visuresp system : wireless inductance plethysmography system

SUMMARY:
Determing optimal time of ventilator disconnection is a challenge for both acute and chronic neuromuscular disease. In one case it is helpful for weanning from ventilator and in the other to optimize daytime ventilation in the most severe patients. The investigators propose to validate a new non invasive tool for monitoring respiratroy parameters in neuromuscular patients in both acute and chronic conditions.

DETAILED DESCRIPTION:
Context:

Mechanical ventilation transformed the prognosis of neuromuscular diseases whether for acute or chronic diseases. The available tools to estimate the severity of respiratory insufficiency and indicate or follow the efficiency of mechanical ventilation are based on blood gazes explorations, tests respiratory function and sleep evaluation.

These tools give either limited information, or are with difficulty applicable to patients heavily handicapped except during hospitalization.

In patients under mechanical ventilation, it is sometimes difficult to know the daily optimal time of ventilation. The respiratory events are not generally recognized and are unspecific (headaches, drowsiness, dyspnoea, etc.) or are identified by blood gazes abnormalities (hypercapnia. In acute setting, treble is going to raise the problem of the weaning of the mechanical ventilation and the optimal moment of the extubation without risking a reintubation.

These problems are identical and concern the evaluation of the degree of ventilatory autonomy for home care. The development of methods estimating this autonomy is thus fundamental.

Objectives: the objective of this project is to validate a non-invasive system for measure and acquisition of respiratory parameters, incorporating a transmission system working by a "wireless" technology allowing the remote monitoring of these patients.

The secondary objectives are to determine the parameters of success of weaning by using the device in neuromuscular patients intubated for respiratory failure in acute setting and to determine the optimal time of free breathing possibilities in patients ventilated in a chronic way at home.

Methods:

After validation of the device on 10 healthy subjects, continuous acquisition of the ventilatory data by means of the Teleresp system compared with measure of the transcutaneous PCO2, of SaO2 and arterial gazometry at the end of free breath trial in 40 acute and chronic neuromuscular patients.

Selection criteria:

Healthy volunteers Patients affected by acute neuromuscular pathology and starting weaning from invasive ventilation (Guillain Barré and myasthenia).

Patients affected by neuromuscular pathology and home ventilated in a diurnal and night-way by invasive interface or not (respiratory autonomy of at least 1:00 am).

Number of patients, center:

10 healthy volunteers and 40 patients hospitalized in the intensive care unit or in the home of ventilation unit of the Raymond Poincaré hospital.

Total duration of the study: 19 months

ELIGIBILITY:
Inclusion Criteria:

Healthy volonteers Man or woman of more than 18 years Realization of a preliminary medical examination Patient having signed an informed and written consent Major healthy subjects, presenting no chronic pathology or not chronic patients

Chronic patients Man or woman of more than 18 years Affected by neuromuscular pathology Realization of a preliminary medical examination Patient in the stable state at the time of the study for at least 1 month Ventilated in a not invasive or invasive way in diurnal and night-period. Respiratory autonomy > 1:00 am Patient having signed an informed and written consent

Acute Patients Man or woman of more than 18 years Affected by syndrome of Guillain blocked in aigue phase having required the invasive ventilation or affected by myasthenia generalized with myasthénique crisis having required the invasive ventilation.

Realization of a preliminary medical examination Patient in phase of neurological recovery Vital Capacity > 15 ml / kg Respiratory Autonomy > 1:00 am Patient having signed a lit(enlightened) and written consent

Exclusion Criteria:

Healthy volonteers subject refusing to participate in the study subject under guardianship or guardianship Pregnant or breast-feeding Woman

Chronic patients Patient refusing to participate in the study Patient under guardianship or guardianship Pregnant or breast-feeding Woman Patients ventilated only at night Clinically significant bronchial Dimensions(Congestion) Required by oxygen therapy

Acute patients Patient refusing to participate in the study Patient or subject under guardianship or guardianship Pregnant or breast-feeding Woman Clinically significant bronchial Dimensions(Congestion) Required by oxygen therapy FIO2 > 40 % PEP > 5 cms H2O State of shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-11; Primary Completion 2012-11 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of pathological respiratory events (apneas, hypopneas, paradoxical breath) detected with regard to the recording of the PtCO2 and the SpO2 | 1 to 12 hours
  Healthy subjects will be recorded for one hour in seated positions 30 minutes and slept 30 min.
  Pneumotachograph recording will be realized during 5 minutes at the beginning and at the end of every phase of recording. The computer assuring the reception of the signals being remotely located to estimate of the transmission.
  All the patients will be registered in parallel with the VISURESP ® system (RBI Grenoble, France) and the measure of the transcutaneous PCO2 and SpO2(SenTec AG, Therwil, Switzerland) during free breath. The measure beginning 30 minutes before the logout and finishing 30 minutes later.
  Acute patients being able to like at least 2 H of free breath will be recorded. A first measure will be made dice that a free breath of at least 2H will be possible, then 3 days later and the day the extubation. Aterial blood gazes will be obtained before reconnection. Chronic patients willbe recorded if able to be disconnected from ventilator for more than 1 hour.

SECONDARY OUTCOMES:
Respiratory events in healthy volonteers | 1h
  Quality of data transmission of respiratory paramaters
Respiratory events in chronic Patients | 1-12h
  Correlation between the number of event detected by VISURESP ®, the duration of hypercapnie superior to 45 mmHg on the PtCO2 and the gazométrie at the end of free Breath.
Respiratory events in acute patients | 1-12h
  Correlations between the number of events detected by the technology VISURESP ®, the duration of hypercapnie superior to 45 mmHg on the PtCO2 and the success of the extubation (at least 24 a hour)

CONTACTS AND LOCATIONS:
Overall Officials: DAVID ORLIKOWSKI, MDPHD, Principal Investigator — Cic it 805
Locations (1):
- Hopital Raymond Poincare, Garches, Île-de-France Region, France

REFERENCES:
- [Background] Modalités pratiques de la ventialtion non invasive en pression positive, au long cours, a domicile, dans les maladies neuromusculaires. Rev Mal Respir 2006;23:S3-S40. Toussaint M, Steens M, Wasteels G, Soudon P. Diurnal ventilation via mouthpiece: survival in end-stage Duchenne patients. Eur Respir J 2006;28(3):549-55. Seneviratne J, Mandrekar J, Wijdicks EF, Rabinstein AA. Predictors of extubation failure in myasthenic crisis. Arch Neurol 2008;65(7):929-33. Prigent H, Orlikowski D, Letilly N, Falaize L, Annane D, Sharshar T, et al. Vital Capacity Versus Maximal Inspiratory Pressure in Patients with Guillain-Barre Syndrome and Myasthenia Gravis. Neurocrit Care. Kohler M, Clarenbach CF, Bahler C, Brack T, Russi EW, Bloch KE. Disability and survival in Duchenne muscular dystrophy. J Neurol Neurosurg Psychiatry 2009;80(3):320-5. Brouillette RT, Morrow AS, Weese-Mayer DE, Hunt CE. Comparison of respiratory inductive plethysmography and thoracic impedance for apnea monitoring. J Pediatr 1987;111(3):377-83. Calabrese P, Besleaga T, Eberhard A, Vovc V, Baconnier P. Respiratory inductance plethysmography is suitable for voluntary hyperventilation test. Conf Proc IEEE Eng Med Biol Soc 2007;2007:1055-7. Eberhard A, Calabrese P, Baconnier P, Benchetrit G. Comparison between the respiratory inductance plethysmography signal derivative and the airflow signal. Adv Exp Med Biol 2001;499:489-94. Redline S, Budhiraja R, Kapur V, Marcus CL, Mateika JH, Mehra R, et al. The scoring of respiratory events in sleep: reliability and validity. J Clin Sleep Med 2007;3(2):169-200.